CLINICAL TRIAL: NCT03596333
Title: Use of Color Doppler Ultrasonography to Confirm the Position of a Labor Epidural Needle - a Retrospective Case Series
Brief Title: Color Doppler Ultrasound to Locate Needle in Labor Epidural
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Other Study IDs: 1230080
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Labor Pain; Obstetric Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective chart review — We conducted a retrospective chart review to evaluate the stored ultrasound images used during labor epidural placement, as well as demographic and anesthetic variables.

SUMMARY:
Color Flow Doppler (CFD) utilizes Doppler information obtained from signals sent to and received from a transducer. This information is color-encoded and then displayed as color on an overlay of the two-dimensional image. The color scale represents both speed and direction of flow within a discrete area of the image. CFD has been recently used to determine the position of the epidural catheter. However its role in labor epidural has yet to be defined. This study describes the use of CFD to confirm the position of the tip of the epidural needle in the context of labor analgesia. This study hypothesized that CFD is a feasible method for identifying proper epidural needle placement prior to epidural catheter advancement.

DETAILED DESCRIPTION:
After obtaining approval by the Institutional Review Board and a waiver of informed consent, thirty-five pregnant patients who underwent an ultrasound guided labor epidural between August of 2017 and June of 2018, were included in this retrospective review. The ultrasound guided labor epidural was used in those in which an anticipated technical difficulty with landmark epidural space localization was expected. These included those patients with diagnosis of obesity and lumbar scoliosis, as well as those with poorly defined surface lumbar bone anatomy. Patients with history of spine surgery were excluded. Patient data were obtained from the institutional electronic medical records. Demographic data, intervertebral level of insertion, dermatome level, and failure rate of epidural needle placement using color flow Doppler were noted for each patient.

Labor analgesia was obtained via a combined spinal epidural technique. Sterile preparation and draping of the area was followed by placement of a curvilinear ultrasound transducer in a sterile sheath. The ultrasound was used to identify the interspinous space. The epidural needle was guided with the use of real time ultrasound by the use of an out of plane technique. A two hand technique was used to manipulate the needle and the ultrasound probe. A 17G Tuohy needle (B. Braun Medical Inc, Bethlhem, PA, USA) was advanced until loss of resistance to normal saline was attained. Confirmation of the epidural space with the use of color flow Doppler (CFD) was then obtained after injection of up to 10 mL of normal saline through the epidural needle. A 27G pencil-point spinal needle (B. Braun Medical Inc, Bethlhem, PA, USA) was then introduced through the epidural needle until cerebro-spinal fluid (CSF) was obtained. Use of intrathecal fentanyl or local anesthetic plus fentanyl was then used as a bolus in the spinal space. A 21G epidural catheter (B. Braun Medical Inc, Bethlhem, PA, USA) was then threaded into the epidural space.

ELIGIBILITY:
Inclusion Criteria:

• Pregnant patients who had labor epidural placed for clinical indications, in whom ultrasound was used to assist the procedure.

Exclusion Criteria:

* Poor quality ultrasound images judged by experienced anesthesiologist
* Patients with history of lumbar spine surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Term pregnant patients who underwent labor epidural assisted with ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Epidural needle tip position | 5 minutes (from insertion of epidural needle until identification of position)
  Identification of posterior complex (dura and ligamentum flavum with color flow Doppler

SECONDARY OUTCOMES:
Epidural catheter position | 5 minutes (from advancement of epidural catheter until identification of position)
  Identification of epidural catheter with color flow Doppler
Epidural failure rate | 12 hours (labor duration)
  Number of failed epidurals requiring replacement

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Riveros Perez, MD, Principal Investigator — Medical College of Georgia. Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided